CLINICAL TRIAL: NCT03953768
Title: Prospective Non-randomized Single-arm Trial of Efferent Neuromodulation Immune and Gastrointestinal Systems by VNS in the Epilepsy Population
Brief Title: VNS Prospective Neuromodulation of Immune and Gastrointestinal Systems
Acronym: VNS-IG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: LivaNova (Industry); Norton Foundation (Unknown)
Responsible Party: Principal Investigator, Ian Mutchnick, Assistant Professor of Neurosurgery, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19.0330
Record Dates: First submitted 2019-04-15; First posted 2019-05-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Diseases; Epilepsy; Autonomic Dysfunction; Inflammatory Bowel Diseases
Keywords: epilepsy; vagal; autoimmune; autonomic; inflammatory bowel disease; immune
MeSH Terms: conditions — Autoimmune Diseases; Epilepsy; Primary Dysautonomias; Inflammatory Bowel Diseases | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective single-arm with internal control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients undergoing device implantation (Experimental): Patients undergoing device implantation with vagal nerve stimulator (VNS) for epilepsy
  Interventions: Device: Vagal nerve stimulation (VNS)

INTERVENTIONS:
Device: Vagal nerve stimulation (VNS) — Implantation with vagal nerve stimulator for epilepsy
  Other Names: Cyberonics VNS

SUMMARY:
Vagal nerve stimulation is a neurosurgical procedure consisting of implantation of an impulse generator battery with leads placed into the vagus nerve in the neck. This procedure was FDA approved for epilepsy in the 1990s and is commonly performed as an outpatient surgery. The mechanism of action is not well understood; however it is increasingly recognized that electrical stimulation of the vagus nerve may impact other organ systems in the body including the immune and gastrointestinal systems. Concrete characterization of the peripheral effects of VNS in human gut microbiome and immune systems will: (1) elucidate peripheral mechanism of action of chronic VNS therapy, (2) identify peripheral preoperative biomarker of VNS efficacy, and (3) create a foundation for research investigating new GM and IM-related disease indications for VNS.

The primary objective of this study is to characterize the pre- and post-operative oral and gut microbiome of patients implanted with vagal nerve stimulator (VNS) for epilepsy. Secondary objectives of this study include: (1) to characterize the pre-operative and post-operative immune profile of patients undergoing VNS implantation for epilepsy, (2) to elucidate whether oral and/or gut microbiota changes are related to VNS efficacy for epilepsy and (3) identification of a biomarker predicting VNS efficacy.

ELIGIBILITY:
Inclusion criteria:

1. Undergoing VNS implantation for the first time as a treatment for epilepsy and
2. Documented follow up with a Louisville-based neurologist in the past 1 year. If at the University of Utah or Baylor University documented ability to travel to their corresponding neurologist.
3. Documented ability to travel to Louisville for outpatient medical care. If at the University of Utah or Baylor University documented ability to travel to their facilities.

Exclusion criteria:

1. Previous treatment with VNS (other than the one implanted for this study)
2. Current pregnancy (contraindication to surgery)
3. Active infection
4. History of cancer or treatment with chemotherapy
5. History of autoimmune disease: Patients who received high effect anticholinergic medication within 30 days of enrollment will be excluded, whereas moderate to low effect anticholinergic medication will be discussed with and decided by the PI.
6. If any high effect anticholinergic medication is started after enrollment, it will be the PI's decision to drop or postpone the corresponding visit or exclude the patient entirely.
7. Patients who received high effect corticosteroids within 30 days of enrollment will be excluded, whereas moderate to low effect corticosteroids will be discussed with and decided by the PI.
8. If any high effect corticosteroid is started after enrollment, it will be the PI's decision to drop or postpone the corresponding visit or exclude the patient entirely.
9. Treatment with antiarrhythmic or (heart) rate controlling medication,
10. Pre-existing cardiac arrhythmia or presence of cardiac pacemaker / defibrillator

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-13 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Metagenomic microbiome profile | 1 year
  Stool and saliva specimens will be used to generate metagenomic profiles of gut flora populations. Pre- and post-VNS gut profiles will be compared. It is important to note that the genomic profile of all gut flora is the outcome, rather than the presence or absence of any specific type of bacteria.
Bowel movement frequency | 1 year
  A brief clinical questionnaire regarding the frequency and consistency of bowel movements will be administered. This will be done pre- and post-VNS implantation in each patient. Any medications to manage diarrhea and constipation will be carefully recorded as well as their efficacy.
Bowel habits | 1 year
  A clinical bowel habits questionnaire will be administered at each study visit to determine changes in bowel habits pre and post operatively. Additionally, the Bristol stool scale will be assessed at each visit.
Immune Profile 1 - Flow cytometric profiling of cell populations | 1 year
  One milliliter of whole blood from each subject will be aliquoted into separate tube and directly stained with fluorochrome-conjugated antibodies to investigate the cellular composition of the blood. Subtypes of lymphocytes, monocytes and granulocytes will be defined by set phenotypic marker expression
Immune Profile 2 - Ex vivo stimulation of cells in whole blood | 1 year
  Up to 10 ml of the whole blood will be cultured in 24-well tissue culture plates in the presence and absence of innate immune cell activators, such as TLR ligands, LPS, CpG ODN, poly I:C or flagellin, or adaptive immune activators such as anti-CD3/anti-CD28 beads, PHA or recall antigens. Culture supernatants and cells will be harvested at the needed time points and analyzed via MSD and qPCR, respectively.
Inflammatory Profile 1 - Meso Scale Discovery (or MSD) analysis for pro-inflammatory cytokines/chemokines | 1 year
  Serum electrochemiluminescence detection analysis of the following cytokines/chemokines: IFNg, IL-1ß, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNFα. Units in Picograms/ml or Nanograms/ml depending on the specific chemokine/cytokine
Inflammatory Profile 2 - Meso Scale Discovery (or MSD) analysis for metabolic hormones | 1 year
  Serum electrochemiluminescence detection analysis of the following hormones: GLP-1, insulin, Glucagon, Leptin. All in picograms/mL.
Inflammatory Profile 3 - Metabolomics for Short Chain Fatty acids (SCFAs) | 1 year
  Short Chain Fatty Acids (SCFAs) in both feces and serum will be derivatized, extracted in organic solvent and analyzed using Gas chromatography-mass spectrometry (GC-MS) to determine the levels of short-chain fatty acids. To the microbial community SCFAs are a necessary waste product, required to balance redox equivalent production in the anaerobic environment of the gut. SCFAs are saturated aliphatic organic acids that consist of one to six carbons of which acetate (C2), propionate (C3), and butyrate (C4) are the most abundant (≥95%). Acetate, propionate, and butyrate are present in an approximate molar ratio of 60:20:20 and will be measured in picomoles/mL.
Inflammatory Profile 4 - Intestinal inflammation and permeability markers | 1 year
  sCD163 (nanograms/mL), sCD14 (micrograms/mL), CRP (mg/L), and I-FABP (picograms/mL) are markers of intestinal inflammation and permeability and will be measured using an enzyme-linked immunosorbent assay (ELISA) performed on cell-free supernatants such as plasma, serum and urine. The units of measurement

SECONDARY OUTCOMES:
Epilepsy severity | 1 year
  Patients will keep a log of seizure type, keeping careful track of the frequency of each type, how long each seizure lasts and what medical interventions are taken to stop each seizure. Additionally, 1 year Engel outcome will be assessed.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No